CLINICAL TRIAL: NCT05030090
Title: Integrative Nutrition Care Plan for the Patient With Liver and Colorectal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Collaborators: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N202105003
Record Dates: First submitted 2021-06-25; First posted 2021-09-01 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2021-06

CONDITIONS: Malnutrition; Cancer of Colon; Cancer of Liver; Nutrition Aspect of Cancer
Keywords: Nutrition care of cancer; Liver cancer; Colorectal cancer; Remote consultation; Nutrition supplement
MeSH Terms: conditions — Malnutrition; Colonic Neoplasms; Liver Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Active Comparator): 1. Consulted by the dietitian using communication software (Line) or telephone.
  2. At 0.5, 1, 1.5, 2, 2.5, and 3 months will track the biochemical data, assess nutritional status and quality of life.
  3. The nutrition care plan period will be three months.
  Interventions: Behavioral: Nutritional consultant
- Nutrition care plan group A (Experimental): 1. Consulted by the dietitian using communication software (Line) or telephone.
  2. Implement a daily diet with a concentrated high-calorie and high-protein liquid supplement
  3. At 0.5, 1, 1.5, 2, 2.5, and 3 months will track the biochemical data, assess nutritional status and quality of life.
  3.The nutrition care plan period will be three months.
  Interventions: Behavioral: Nutritional consultant; Dietary Supplement: Nutritional consultant + High-calorie, high-protein liquid nutrition supplement
- Nutrition care plan group B (Experimental): 1. Consulted by the dietitian using communication software (Line) or telephone.
  2. Implement a daily diet with a concentrated high-calorie and high-protein liquid supplement and powdered supplement 1 and nutritional products and powdered supplement 2
  3. At 0.5, 1, 1.5, 2, 2.5, and 3 months will track the biochemical data, assess nutritional status and quality of life.
  4. The nutrition care plan period will be three months.
  Interventions: Behavioral: Nutritional consultant; Combination Product: Nutritional consultant + Liquid supplement + Powdered supplement 1 and 2

INTERVENTIONS:
Behavioral: Nutritional consultant — The control group is to be consulted by the dietitian using communication software (Line) or telephone to evaluate the nutritional requirement and guide the cancer diet principles before starting the project.
Dietary Supplement: Nutritional consultant + High-calorie, high-protein liquid nutrition supplement — At the beginning of the plan, the dietitian first calculates the patient's daily calorie intake and the ratio of the three macronutrients and guides the patients or their family members of the nutritional care plan group A to implement a daily diet with a concentrated high-calorie and high-protein liquid supplement (Commercial formula contains 425 kcal and 19.1 grams of protein).
  Arms: Nutrition care plan group A
Combination Product: Nutritional consultant + Liquid supplement + Powdered supplement 1 and 2 — At the beginning of the plan, the dietitian first calculates the patient's daily calorie intake and the ratio of the three macronutrients and guides the patients or their family members of the nutritional care plan group B to implement a daily diet with a concentrated high-calorie and high-protein liquid supplement (Commercial formula contains 425 kcal and 19.1 grams of protein). Meanwhile, nutrition care plan group B will be given powdered supplement 1 (containing β-glucan and gamma-aminobutyric acid) and nutritional products and powdered supplement 2 (contains water-soluble dietary fiber and probiotics).
  Arms: Nutrition care plan group B

SUMMARY:
At present, the families of cancer patients are lack knowledge and experience of nutritional care after discharge. As a result, cancer patients often suffer from low nutritional status after being discharged from the hospital.

DETAILED DESCRIPTION:
This study intends to design a home nutrition care plan to explore the effect of a home nutrition care plan on the nutritional status of patients with liver cancer and colorectal cancer at risk of malnutrition. Malnutrition or side effects often lead to natural food intake for patients. It is not enough to meet the nutritional requirements, so it is matched with dietary products to help patients more easily meet their nutritional requirements. Supplements are used to alleviate patients' side effects. It is hoped that they can help patients improve their nutritional status.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with liver cancer or colorectal cancer stage I to III
2. Not suffering from other carcinomas in situ at the same time
3. Will undergo surgery or non-surgical cancer treatment
4. Can move, read and answer questions by itself
5. At least one social support (family or friend) to assist and support the patient to complete the trial
6. According to the aPG-SGA, the assessment score is between 4 ~ 9
7. The patient or caregiver can cooperate with the dietitian to track and answer related questions asked by the dietitian in a remote way through communication software or telephone every week.
8. Able to adjust diet or take nutrition and supplements daily with the guidance of a nutritionist
9. Be able to cooperate with doctors and the beginning of the study and monthly return visits and blood tests for health insurance items

Exclusion Criteria:

1. Perform organ transplantation or palliative care
2. Hepatic encephalopathy
3. History of cardiovascular and cerebrovascular diseases
4. Severe organ failure of the heart, breathing, or kidneys
5. History of digestive tract inflammation or ulcer
6. Severe mental illness
7. An active infectious diseases
8. Those who can only use intravenous nutrition and cannot use enteral nutrition
9. People who are allergic to product ingredients (milk, soy, or mango and their products)
10. Unwilling to cooperate with dietitians to make dietary adjustments or supplement nutrition and supplements
11. Unwilling to actively treat cancer

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2021-06-25 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Evaluate nutritional status indicators change | Baseline and at 0.5th month
  Improvement of nutritional status indicators: Abridged Patient-Generated Subjective Global Assessment (aPG-SGA) assessment scores.
Evaluate nutritional status indicators change | Baseline and at 1st month
  Improvement of nutritional status indicators: Abridged Patient-Generated Subjective Global Assessment (aPG-SGA) assessment scores.
Evaluate nutritional status indicators change | Baseline and at 1.5th month
  Improvement of nutritional status indicators: Abridged Patient-Generated Subjective Global Assessment (aPG-SGA) assessment scores.
Evaluate nutritional status indicators change | Baseline and at 2nd month
  Improvement of nutritional status indicators: Abridged Patient-Generated Subjective Global Assessment (aPG-SGA) assessment scores.
Evaluate nutritional status indicators change | Baseline and at 2.5th month
  Improvement of nutritional status indicators: Abridged Patient-Generated Subjective Global Assessment (aPG-SGA) assessment scores.
Evaluate nutritional status indicators change | Baseline and at third month
  Improvement of nutritional status indicators: Abridged Patient-Generated Subjective Global Assessment (aPG-SGA) assessment scores.

SECONDARY OUTCOMES:
Evaluate anthropometric measurements change-Body weight | Baseline and at 0.5th, 1st, 1.5th, 2nd, 2.5th, and third month
  Weight in kilograms
Evaluate anthropometric measurements change-Body mass index(BMI) | Baseline and at 0.5th, 1st, 1.5th, 2nd, 2.5th, and third month
  Weight and height will be combined to report BMI in kg/m^2
Evaluate biochemical data change-White blood cells (WBC) | Baseline and at 1st, 2nd, and third month
  White blood cells (x10^3/ul)
Evaluate biochemical data change-Red blood cells (RBC) | Baseline and at 1st, 2nd, and third month
  Red blood cells (x10^6/ul)
Evaluate biochemical data change-Hemoglobin (Hb) | Baseline and at 1st, 2nd, and third month
  Hemoglobin (g/dl)
Evaluate biochemical data change-Hematocrit (Hct) | Baseline and at 1st, 2nd, and third month
  Hematocrit (%)
Evaluate biochemical data change-Platelet | Baseline and at 1st, 2nd, and third month
  Platelet (x10^3/ul)
Evaluate biochemical data change-Mean corpuscular volume (MCV) | Baseline and at 1st, 2nd, and third month
  Mean corpuscular volume (fl)
Evaluate biochemical data change-Mean corpuscular hemoglobin (MCH) | Baseline and at 1st, 2nd, and third month
  Mean corpuscular hemoglobin (pg)
Evaluate biochemical data change-Mean corpuscular hemoglobin concentration (MCHC) | Baseline and at 1st, 2nd, and third month
  Mean corpuscular hemoglobin concentration (g/dl)
Evaluate biochemical data change-Neutrophil band | Baseline and at 1st, 2nd, and third month
  Neutrophils (%), Lymphocyte (%), Monocyte (%), Eosinophil (%), and Basophil (%)
Evaluate biochemical data change-renal function | Baseline and at 1st, 2nd, and third month
  Blood urea nitrogen and Creatinine (mg/dl)
Evaluate biochemical data change-Albumin (Alb) | Baseline and at 1st, 2nd, and third month
  Albumin (g/dl)
Evaluate biochemical data change-liver function | Baseline and at 1st, 2nd, and third month
  Aspartate aminotransferase and Alanine aminotransferase (U/l)
Evaluate biochemical data change-renal function | Baseline and at 1st, 2nd, and third month
  estimated Glomerular filtration rate (eGFR) (mL/min/1.73 m^2)
Evaluate biochemical data change-lipid profile | Baseline and third month
  Triglyceride, Total cholesterol, Low-density lipoprotein cholesterol, High-density lipoprotein cholesterol (mg/dl)
Evaluate food intake change (energy) | Baseline and at 0.5th, 1st, 1.5th, 2nd, 2.5th, and third month
  Use 24-hour dietary recall to evaluate the nutrition intake (energy in calories)
Evaluate food intake change (protein) | Baseline and at 0.5th, 1st, 1.5th, 2nd, 2.5th, and third month
  Use 24-hour dietary recall to evaluate the nutrition intake (protein in grams)
Evaluate quality of life indicators change | Baseline and at 0.5th, 1st, 1.5th, 2nd, 2.5th, and third month
  Scores on the Quality of Life Scale (European Organization for Research and Treatment of Cancer quality of life questionnaires core 30, EORTC QLQ-C30)

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Medical University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No